CLINICAL TRIAL: NCT04098341
Title: Uptake, Effectiveness and Acceptability of Routine Screening of Pregnant Migrants for Latent Tuberculosis Infection in Antenatal Care: a Feasibility Study
Brief Title: Screening for Tuberculosis in Pregnancy
Acronym: STOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: University College, London (Other); City, University of London (Other); Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRAS247388 REC19/LO/0557
Record Dates: First submitted 2019-08-05; First posted 2019-09-23 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Latent Tuberculosis
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Intervention Model Description: Observational study assessing the feasibility and acceptability of opt-out screening for latent Tuberculosis infection amongst pregnant migrants in antenatal clinics. All pregnant migrants who meet the inclusion criteria will be offered an opt-out IGRA blood test as screening for latent TB infection
Masking Description: as above
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening (Other): All eligible migrants will be offered opt-out IGRA blood test to screen for for latent Tuberculosis infection
  Interventions: Diagnostic Test: IGRA blood test used as a tool for opt-out screening for latent Tuberculsis infection

INTERVENTIONS:
Diagnostic Test: IGRA blood test used as a tool for opt-out screening for latent Tuberculsis infection — All eligible pregnant migrants will be offered an opt-out screening IGRA blood test for latent Tuberculosis infection

SUMMARY:
The UK has the second highest tuberculosis (TB) incidence in Western Europe. Most active cases occur in migrants due to reactivation of latent TB infection (LTBI) acquired abroad. Screening migrants for LTBI was recently introduced by Public Health England to reduce TB rates and transmission of infectious cases. Newham, which has one of the highest TB rates in London introduced the first large-scale LTBI screening programme for migrants, but it is poorly accessed by pregnant women and screening uptake is low. The issue of how best to screen for TB during pregnancy is important because pregnant/ postpartum women are at particularly high risk of developing TB, and migrants from countries with high TB rates may only interact with healthcare services during pregnancy.

Effective strategies are urgently needed to improve screening uptake for LTBI in pregnant migrants. The Antenatal clinic is an attractive location to screen for LTBI because uptake and acceptability of opt-out screening for other infectious diseases (HIV) is high. We will evaluate the uptake, effectiveness and acceptability of routine screening for LTBI in antenatal clinics. Eligible patients are pregnant women who have entered the UK within 10 years from a country with TB rates of >150/100,000. Screening will involve a blood test, taken with other routine antenatal blood tests. We expect that in this setting, screening will be acceptable and uptake will be high. Our main outcome will be to assess the uptake of screening in at least 200 women. Acceptability of screening and understanding barriers of healthcare professionals to test for LTBI are secondary aims. The study will provide important information about a new setting in which to screen pregnant migrants for LTBI and barriers to starting treatment postpartum, which will inform the definitive trial to guide national policy on LTBI screening in antenatal care.

DETAILED DESCRIPTION:
The UK has the second-highest TB incidence in Western Europe. Most active TB cases occur in the non-UK born population (migrants) in large cities such as London. Migrants most at risk of TB are from countries with a high TB incidence such as the Indian subcontinent and Sub-Saharan Africa. One quarter of the whole world population are estimated to have LTBI. Migrants who have acquired LTBI outside the UK, often reactivate in the first 5-10 years after arrival. Barts Health NHS trust has one of the highest number of TB notifications in England and manages 8% of active TB cases in the UK.

Many countries in SE Asia and Africa, which have the highest global TB burden, also have high maternal mortality rates. In women of reproductive age (15-45 years), TB is now among the three leading causes of death. In 2014, an estimated 480,000 women died as a result of TB globally. TB diagnosis in pregnancy is often delayed even in low-incidence countries. Pregnancy can mask the clinical manifestations of TB, as some of the symptoms of TB such as fatigue and loss of appetite are also common in pregnancy itself. There is a high risk of LTBI reactivation during pregnancy and postpartum likely due to T-cell suppression and reduced interferon-gamma production.There is an elevated risk of TB during pregnancy and immediately postpartum compared to the general population. TB in pregnancy carries a high risk of perinatal complications, poor foetal and maternal outcomes and early diagnosis of TB is important to prevent significant maternal and perinatal complications. A simple clinical algorithm recommended by the WHO based on absence of current cough, fever, weight loss, and night sweats can help to exclude active TB disease. Sputum smear has a low sensitivity for diagnosis of active TB in pregnancy, however health care professionals will have a higher index of suspicion for active TB in IGRA positive pregnant women presenting with symptoms suggestive of TB, thus preventing a delay in diagnosis. TB diagnosis in pregnancy can be delayed due to reduced awareness among health care providers and reluctance to investigate non-specific TB symptoms by chest radiography. Pregnant migrants may not be accessing routine health care and often do not have a GP. Antenatal care may therefore be a rare and critical opportunity to assess a woman's health and screen for TB. Moreover, antenatal care provides an opportunity for health promotion such as advocating GP registration. England's collaborative TB strategy recommends migrant screening for LTBI in high incidence areas in England including boroughs such as Newham. LTBI screening programmes have now been implemented. Between April 2015 and June 2016, 5,622 eligible migrants in England were offered an LTBI test, 2,904 (51%) of whom attended for the test. Newham was the first London borough to introduce a large-scale LTBI screening programme. A total of 20,905 LTBI tests were reported between July 2014 and June 2017 across England, nearly half of the tests were reported in Newham however uptake of screening remains low. This may be because individuals eligible for screening do not have symptoms and perceive the risk of developing active TB as low. Newham data has shown that uptake of screening varies significantly amongst GP surgeries indicating that uptake may be influenced by healthcare providers' knowledge and attitudes to screening but may also be due to other factors such as proximity to phlebotomy services. Data from the Clinical Effectiveness Group (CEG) at QMUL has shown that in pregnant migrant women screening uptake is even lower, <25% and this may be because pregnant women have not been told that LTBI screening is important. There is limited qualitative research about the acceptability to women of LTBI screening in pregnancy. Reasons for low uptake may be due to stigma of having active TB or fear of a positive test result affecting their immigration status. An opt-out approach normalises screening that otherwise may present barriers in relation to stigma.

Provider knowledge and understanding of the risks of TB screening and treatment is a major predictor of successful management of TB. Newham data has shown that offer of screening varies significantly amongst GP surgeries indicating that health care provider knowledge and attitude may influence offer of screening.

Evaluating the impact of healthcare provider training to improve TB management has mainly been performed in low income countries and there are only a few rigorous TB training evaluation studies available. E-learning modules use pre- and post- training tests to evaluate acquired knowledge. A GP E-learning module has been developed by TB Alert to enhance knowledge of GPs responsible for screening and treatment of LTBI but the effectiveness of the module has not been formally evaluated.

Aim of the feasibility study The investigator's aim is to assess whether it is feasible and acceptable to screen an at-risk migrant population for latent tuberculosis infection (LTBI) at routine antenatal booking visits in secondary care, using opt-out Interferon- gamma release assay (IGRA) testing. This will allow the investigators to develop a definitive large scale cluster randomised controlled trial (RCT) to evaluate the effectiveness of acceptable interventions to maximise migrant screening for LTBI in pregnancy, and to increase uptake of LTBI treatment postpartum.

Primary objective:

To obtain

Real time continuous data on study design:

* Numbers and proportions of pregnant migrant women eligible for opt-out screening with an IGRA blood test for LTBI in the antenatal care setting.
* The proportion of eligible women who are offered opt-out LTBI screening by healthcare providers.
* Rate of uptake of the opt-out IGRA blood test screening for LTBI, i.e. the percentage of women offered who have the test performed.

Credible understanding of study process:

* Information on the feasibility and practicality of the data collection for the assessment of LTBI at baseline and subsequent visits.
* The appropriate level of support needed for health care providers at site-level to ensure successful recruitment.

Secondary objective

* Preliminary estimates of disease burden to inform the definitive study
* To identify the characteristics of pregnant women associated with accepting LTBI screening.
* To estimate the prevalence of active TB and LTBI in the pregnant migrant cohort.
* Assessment of acceptability of opt-out testing and perceptions about screening for LTBI
* To assess participants' perceptions of the TB and LTBI screening process.
* To determine if IGRA testing is an acceptable intervention to be performed using an opt-out approach in antenatal clinics.
* To evaluate facilitators and barriers to the uptake of LTBI screening among pregnant migrant women and to identify what type of intervention might be effective in increasing awareness.
* To assess participants' perception of the risks and benefits of LTBI screening, and any LTBI treatment, to themselves and their babies.
* To assess participants' perceptions of the timing of treatment (during pregnancy, post-delivery or after termination of breast feeding).
* To understand health care providers' experiences of the screening process and perceived barriers and facilitators to screening uptake.
* To assess participants and heath care providers views on implementation of interventions such as text messaging to increase uptake of LTBI screening and treatment.

To develop acceptable interventions to increase TB awareness among pregnant migrants and health care providers, thereby increasing uptake of screening, such as

* Educational materials or approaches co-developed with TB Alert to increase knowledge about signs and symptoms of TB among pregnant migrant women.
* E-learning modules for midwives and other health care providers to increase knowledge about TB and LTBI.

To collect relevant cost data to assess the cost- effectiveness of LTBI screening in antenatal care compared to screening in primary care in future definitive trial.

• To test the feasibility of collecting cost data

Definitive trial objectives Primary objective

• To evaluate the effectiveness of interventions to increase uptake of migrant screening for LTBI in pregnancy

Secondary objectives

* To study the effectiveness of interventions to increase uptake of LTBI treatment postpartum.
* To evaluate the safety and timing of LTBI treatment postpartum - immediately postpartum or after cessation of breast feeding
* To determine cost-effectiveness of LTBI screening in antenatal care by preventing cases of active TB.

Study design

Consent Posters will be displayed in antenatal clinics explaining the study. All patients will be given a Patient Information Sheet by their midwives that explains the study and what participation will entail.

Valid implied consent will be used for participation in the study and data collection. Written informed consent will be taken for LTBI questionnaires, interviews and focus groups. Furthermore written informed consent will be obtained for questionnaires, knowledge quiz, interviews and focus groups from healthcare providers participating in the study.

Data collection Basic data on age, ethnicity, socioeconomic status, and substance misuse and pre-existing medical conditions (such as diabetes) and antenatal history and TB history will be recorded in all patients electronically in antenatal care according to existing protocols as part of standard of care.

Setting Antenatal clinics at Royal London Hospital, Whipps Cross University Hospital and Newham University Hospital.

Planned intervention

Study Intervention All women who are eligible for LTBI screening and attend the antenatal clinic for their dating scan will be asked to be tested for LTBI alongside other routine investigations for blood borne viruses. IGRA testing will be offered on an opt-out basis similar to HIV testing. In addition, all migrants will be screened for active TB by their midwives using a standardized symptom assessment questionnaire that includes the WHO recommended TB symptom screen. TB awareness-raising will be delivered in antenatal clinics by midwives, utilizing evidence-based tools created by TB Alert. Pregnant women will also be asked to complete a short questionnaire on acceptability of LTBI screening, knowledge about TB/LTBI, and barriers to screening. At the end of pregnancy, women will be asked again to complete a questionnaire to compare the perception and knowledge of active TB/LTBI before and after the screening intervention.

Pregnant women with LTBI will be closely monitored for active TB during pregnancy by their midwives. The GP will be informed of a positive IGRA test and also the TB clinic will be notified. The GP will be asked to refer the patient to TB clinic for LTBI treatment or if the woman lives in Newham she will be treated in primary care. In case this does not happen, the TB clinic will send a reminder to the GP to refer the patient. If women develop symptoms of active TB, the midwife will arrange referral to the TB clinic.

Health care providers involved in antenatal care will be asked to complete an E-learning module on active TB/ LTBI which will be developed by TB Alert and the Royal College of Midwives. The E-learning course, which will be CPD accredited, has a pre and post-course quiz to assess any change in knowledge. Health care providers will be also asked to take part in interviews, focus groups and to complete a questionnaire for which the investigators will obtain written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant migrants aged 16-35 who have entered the UK less than 5 years ago from a country with a TB incidence of greater than 150/100,000 or sub-Saharan Africa

Exclusion Criteria:

* Patients who do not meet the criteria for LTBI screening will be excluded which include:

  1. Previous history of TB or LTBI.
  2. Individuals who are unable to consent.
  3. Evidence of active TB (based on history, examination, blood tests, chest X-ray finding or other radiological findings).

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — biological females who are pregnant
Enrollment: 310 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Uptake of screening for LTBI in antenatal care assessed by calculating the percentage of patients who accepted LTBI screening. | 12 months
  as above
Offer of IGRA blood test screening by healthcare providers assessed by the percentage of eligible women who were offered a test. | 12 months
  as above
Process outcomes for the feasibility study | 21 months
  Proportion of eligible women who are screened, all pregnant women booked for antenatal care will be screened if fulfilling the eligibility criteria, and we will monitor the reasons for ineligibility.

SECONDARY OUTCOMES:
Disease related outcomes | 12 months
  Rates of LTBI prevalence in the pregnant migrant population as assessed by the proportion of IGRA positive migrants.
Disease related outcomes | 12 months
  Rates of active TB identified in pregnant migrants during the study period and time to diagnosis.
Acceptability outcomes | 18 months
  Acceptability of interventions such as educational material to increase uptake of LTBI screening assessed by interviews and focus groups.
Acceptability outcomes | 18 months
  Acceptability of LTBI screening (Perceptions, barriers and facilitators) among pregnant women assessed by qualitative methods (interviews, focus groups) and a standardised non-validated questionnaire.
Acceptability outcomes | 18 months
  Acceptability of treatment for LTBI postpartum and timing of treatment as assessed by interviews and focus groups.
Acceptability outcomes | 18 months
  Identification of barriers influencing uptake of LTBI treatment of migrant women postpartum assessed by interviews and focus groups
Acceptability outcomes | 18 months
  Acceptability of interventions to increase LTBI treatment postpartum such as SMS messaging assessed by interviews and focus groups.
Acceptability outcomes | 18 months
  Acceptability of LTBI screening from a health care providers' perspective assessed by interviews and focus groups.
Knowledge of disease related outcomes | 18months
  Standardised non-validated LTBI knowledge questionnaires at the beginning of pregnancy and after delivery to assess change in knowledge and awareness about active TB/ LTBI amongst migrant women.
Knowledge of disease related outcomes | 18months
  Change in knowledge and awareness about active TB/LTBI amongst healthcare providers assessed by a quiz at the beginning and end of the study evaluating the knowledge gained through the E-learning module and educational programme.
Cost effectiveness outcomes | 21 months
  Calculated as total cost of offering IGRA in antenatal care and comparing it to total cost of offering IGRA in primary care.

CONTACTS AND LOCATIONS:
Overall Officials: Heinke Kunst, Principal Investigator — Queen Mary University of London (study chief investigator)
Locations (3):
- United Kingdom (3):
  - Royal London Hospital, London, Essex
  - Whipps Cross Hospital, London, Essex
  - Newham University Hospital, London, Essex

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahman A, Thangaratinam S, Copas A, Zenner D, White PJ, Griffiths C, Abubakar I, McCourt C, Kunst H. A feasibility study evaluating the uptake, effectiveness and acceptability of routine screening of pregnant migrants for latent tuberculosis infection in antenatal care: a research protocol. BMJ Open. 2022 Apr 4;12(4):e058734. doi: 10.1136/bmjopen-2021-058734. PMID 35379641